CLINICAL TRIAL: NCT02096224
Title: Comparison of the Effects of Sevoflurane and Desflurane on Prevention of Catheter-related Bladder Discomfort
Brief Title: Sevoflurane Versus Desflurane for Catheter-related Bladder Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRBDSevoDes
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-03

CONDITIONS: Catheter Site Discomfort; Complications; Anesthesia; Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Experimental): Sevoflurane will be administered as the maintenance agent of general anesthesia.
  Interventions: Drug: Sevoflurane
- Desflurane (Active Comparator): Desflurane will be administered as the maintenance agent of general anesthesia.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane will be used.
  Arms: Sevoflurane
Drug: Desflurane — Desflurane will be used
  Arms: Desflurane

SUMMARY:
We want to evaluate the efficacy of the sevoflurane and desflurane for the prevention of catheter-related bladder discomfort.

DETAILED DESCRIPTION:
The mechanism of catheter-related bladder discomfort is thought to be related to the muscarinic receptor. The volatile anesthetics such as sevoflurane and desflurane are known to block the muscarinic receptor in different ways.

We want to evaluate the efficacy of the sevoflurane and desflurane for the prevention of catheter-related bladder discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for transurethral bladder excision under general anesthesia
* ASA I-III

Exclusion Criteria:

* Bladder outflow obstruction
* Overactive bladder
* End-stage renal disease
* Neurogenic bladder
* Heart failure
* Arrhythmia
* Morbid obesity
* Use of chronic analgesic medication
* Hepatic disease
* Pulmonary disease
* Psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Catheter-related bladder discomfort | 24 hour postoperatively
  Catheter-related bladder discomfort will be measured for 24 hour postoperatively (0:none, 1:mild, 2:moderate, 3:severe).

SECONDARY OUTCOMES:
Catheter-related bladder discomfort | 0, 1, 6 and 24 hour postoperatively
  Catheter-related bladder discomfort will be measured at 0, 1, 6 and 24 hour postoperatively (0:none, 1:mild, 2:moderate, 3:severe).
Nausea | 0, 1, 6 and 24 hour postoperatively
  The degree of nausea will be assessed as none, mild, moderate and severe at 0, 1, 6 and 24 hour postoperatively.
Vomiting | 0, 1, 6 and 24 hour postoperatively
  The degree of vomiting will be assessed as none, mild, moderate and severe at 0, 1, 6 and 24 hour postoperatively.
Dry mouth | 0 houe after admission of operating room
  Dry mouth after the admission of operating room will be assessed. (score:0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyoung Park, PhD, Study Chair — Seoul National University of Hospital
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HC, Hong WP, Lim YJ, Park HP. The effect of sevoflurane versus desflurane on postoperative catheter-related bladder discomfort in patients undergoing transurethral excision of a bladder tumour: a randomized controlled trial. Can J Anaesth. 2016 May;63(5):596-602. doi: 10.1007/s12630-016-0600-7. Epub 2016 Feb 1. PMID 26830645